CLINICAL TRIAL: NCT04723342
Title: Treatment of Children and Adolescents With Primary B-precursor Acute Lymphoblastic Leukemia With Combination Chemotherapy and Immunotherapy
Brief Title: Acute Lymphoblastic Leukemia Treatment Protocol Moscow-Berlin 2019 Pilot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal Research Institute of Pediatric Hematology, Oncology and Immunology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALL-MB 2019 Pilot
Record Dates: First submitted 2021-01-19; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Childhood Acute Lymphoblastic Leukemia
Keywords: Acute lymphoblastic leukemia; Children; Chemotherapy; Immunotherapy; Blinatumomab
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blinatumomab (Experimental): Consolidation therapy with Blinatumomab administration
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab, intravenously, as continuous 24 hours infusion 1-7 days - 5 μg/m2/day, 8-28 day - 15 μg/m2/day
  1 course after induction treatment

SUMMARY:
THE PURPOSE OF THE STUDY is to optimize the therapy of patients with primary B-cell precursor acute lymphoblastic leukemia (BCP-ALL) by including monoclonal bispecific antibodies in post-induction treatment with simultaneous reduction of chemotherapy.

QUESTIONS AND OBJECTIVES OF THE STUDY:

* to determine the efficacy and feasibility of chemotherapy and immunotherapy combination in comparison with standard PCT in children and adolescents with newly diagnosed BCP-ALL;
* to determine the safety and toxicity of chemotherapy and immunotherapy combination in comparison with standard PCT in children and adolescents with newly diagnosed BCP-ALL;
* to determine the possibility of chemotherapy reducing when immunotherapy is included in the treatment regimen without loss of effectiveness;
* to determine the possibility of reducing the maintenance therapy duration to 1 year when immunotherapy is included in the treatment regimen without loss of effectiveness.

ELIGIBILITY:
Inclusion Criteria:

This study included patients with B-cell precursor ALL (BCP-ALL) diagnosed or confirmed in one of the clinics participating in the study. Also following criteria should be considered at the diagnosis for each case:

1. Age at diagnosis at 1 to 18 years.
2. The start of induction therapy within a time interval of study recruitment phase.
3. The diagnosis of BCP-ALL is to be proved by the morphological, cytochemical, and immunological analysis of tumor cells in bone marrow in the reference laboratories of Dmitry Rogachev National Medical Research Center of Pediatric Hematology, Oncology and Immunology (D. Rogachev NMRCPHOI).
4. CD19 expression on tumor cells.
5. Informed consent of the patient parents (guardians)

Exclusion Criteria:

1. Any non-compliance with the inclusion criteria.
2. ALL is a second malignancy.
3. There is severe concomitant disease, which significantly impedes chemotherapy protocol (such as multiple malformations, heart diseases, metabolic disorders, etc.);
4. The patient was treated before for a long time with cytotoxic drugs.
5. Initial CNS (central nervous system) involvement (status CNSII or CNSIII).
6. Initial leukocyte count ≥100×109/L (except for patients with significant translocations).
7. Patients not achieved cytological remission after induction

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease level | On the last day of the blinatumomab course, on average at 11 weeks of protocol
Minimal residual disease level | 6 months after starting maintenance therapy
Minimal residual disease level | 1 year after starting maintenance therapy
Event-free survival | 3 years after study start
Event-free survival | 5 years after study start

SECONDARY OUTCOMES:
Overall survival | 3 years after study start
Overall survival | 5 years after study start
Cumulative incidence of relapse | 3 years after study start
Cumulative incidence of relapse | 5 years after study start
Remission death rate | 3 years after study start
Remission death rate | 5 years after study start

CONTACTS AND LOCATIONS:
Overall Officials: Alexander I. Karachunskiy, Professor,MD, Principal Investigator — Federal Research Institute of Pediatric Hematology, Oncology and Immunology
Locations (4):
- Russia (4):
  - Dmitry Rogachev National Medical Research Centre of Pediatric Hematology, Oncology and Immunology, Moscow
  - National Medical Research Center of Oncology named after N.N. Blokhin, Moscow
  - Russian Children's Clinic Hospital; Pirogov Russian National Research Medical University, Moscow
  - Almazov National Medical Research Centre, Saint Petersburg